CLINICAL TRIAL: NCT02739568
Title: Efficacy and Safety of Pitolisant (BF2.649) in the Treatment of Excessive Daytime Sleepiness in Patients With Obstructive Sleep Apnea Syndrome, Treated or Not by Nasal Continuous Positive Airway Pressure, But Still Complaining of Excessive Daytime Sleepiness
Brief Title: Pitolisant (BF2.649) in the Treatment of EDS in Patients With OSA
Acronym: HAROSA3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioprojet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P15 13/ BF2.649
Record Dates: First submitted 2016-03-31; First posted 2016-04-15 (Estimated); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Excessive Daytime Sleepiness; Obstructive Sleep Apnea
Keywords: EDS; OSA
MeSH Terms: conditions — Disorders of Excessive Somnolence; Sleep Apnea, Obstructive | interventions — pitolisant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pitolisant (BF2.6449 (Experimental): Histamine H3 receptor H3R antagonist/ inverse agonist
  Interventions: Drug: Pitolisant (BF2.649)
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pitolisant (BF2.649)
  Arms: Pitolisant (BF2.6449
Drug: Placebo
  Arms: Placebo

SUMMARY:
The first objective of this study is to demonstrate the efficacy and safety of pitolisant given at 10, 20, or 40 mg per day versus placebo during 12 weeks of the Double Blind period, to treat the Excessive Daytime Sleepiness (EDS) in patients with Obstructive Sleep Apnea (OSA) refusing the nasal Continuous Positive Airway Pressure (nCPAP) therapy or treated by nCPAP but still complaining of EDS.

The secondary objectives of the study include assessing the long-term tolerance as well as the maintenance of efficacy of pitolisant given at 10, 20 or 40 mg per day during 39 weeks of Open Label Extension period and further investigating the co-variates or co-medications that affect the pharmacokinetics of pitolisant in the target population.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female outpatients aged from at least 18 years
* Patients complaining of EDS refusing to be treated by nCPAP therapy or having been submitted to nCPAP therapy for a minimum period of 3 months, and still complaining of EDS despite the efforts made beforehand to obtain an efficient nCPAP therapy
* Polysomnography performed (for patients submitted to nCPAP therapy - under nCPAP) between V1 and V2 or during the last 12 months with Apnea-Hypopnea Index (AHI): for patients without nCPAP therapy ≥ 15; for patients under nCPAP therapy less or equal to 10
* For patients submitted to nCPAP therapy: nCPAP ≥ 4 hours / day (compliance checked on the clock-time counter of the CPAP machine)
* Mini Mental State Examination (MMSE) ≥ 28
* Beck Depression Inventory - 13 items (BDI-13) score < 16 and item G (suicidal ideation) of BDI-13 = 0
* Body Mass Index (BMI )less or equal to 40 kg/m²
* Epworth Sleepiness Scale (ESS) ≥ 12
* Female patients with child-bearing potential using a medically accepted method of birth control (i.e. oral contraceptives of normal average dosage) agreeing to continue this method throughout the study, and during the month following treatment discontinuation, being negative to serum pregnancy test performed at the screening visit
* If specified by the investigator, the patient must be willing not to operate a car (if sleepy at wheel) or heavy machinery for the duration of the trial or as long as the investigator deems it clinically indicated. In addition, the patient should be willing to maintain during the study their usual behaviors which could affect their diurnal sleepiness (e.g. circadian rhythm, caffeine consumption, nocturnal sleep duration)
* Patients having signed and dated the informed consent form

Exclusion Criteria:

* Patients suffering from chronic severe insomnia in accordance with the International Classification of Sleep Disorders (ICSD 2005) without OSA
* Patients with co-existing narcolepsy (ICSD 2005), judged on clinical criteria
* Patients with sleep debt not due to OSA (according to the physician' s judgment)
* Patients with non-respiratory sleep fragmentation (restless leg syndrome…)
* Shift work, professional drivers

  * Refusal from the patient to stop any current therapy for EDS or predictable risk for the patient to stop the therapy
  * Patients suffering from a psychiatric disease
  * Acute or chronic disease preventing the improvement assessment, e.g. severe chronic obstructive pulmonary disease (COPD)
  * Current or recent (within one year) history of drug, alcohol, narcotic or other substance abuse or dependence
  * Any significant serious abnormality of the cardiovascular system, e.g. recent myocardial infarction, angina, hypertension or dysrhythmias (within the previous 6 months), Electrocardiogram Fridericia corrected QT interval higher than 450 ms, history of left ventricular hypertrophy or mitral valve prolapse
  * Severe co-morbid medical or biological conditions that may jeopardize study participation at the discretion of the investigator (particularly in the cardiovascular system and the instable diabetes)
  * Positive serology tests (HIV, HCV and HBsAg)
  * Pregnant or breast-feeding women
  * Women with child-bearing potential and no efficient birth-control method
  * Patients unable to understand the study protocol
  * Patients with suspected or known hypersensitivity to study medication
  * Patients with a dominant arm deficiency impeding the achievement of the tests
  * Patients using a prohibited medication
  * Congenital galactose poisoning, glucose and galactose malabsorption, deficit in lactase
  * Patients participating in another study or being in a follow-up period for another study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Epworth sleepiness scale (ESS) | at weeks 12 and 52
  Change from Baseline of ESS

SECONDARY OUTCOMES:
Percentage of ESS responders | at weeks 12 and 52
  Percentage of ESS responders
Reduction of sleepiness and sleep episodes on the sleep diary | at weeks 12 and 52
  Reduction of sleepiness and sleep episodes
Improvement in vigilance according to Oxford Sleep Resistance (OSleR) test | at weeks 12 and 52
  Improvement in vigilance according to Oxford Sleep Resistance (OSleR) test
European Quality of Life Questionnaire (EQ-5D) | at weeks 12 and 52
  EQ-5D improvement (mobility, self-care, usual activities, pain/discomfort and anxiety/depression)
Leeds Sleep Evaluation Questionnaire (LSEQ) | at weeks 12 and 52
  LSEQ improvement (changes in sleep and next morning behaviour during disease/pharmacological investigations)
The Pichot Fatigue Scale | at weeks 12 and 52
  Pichot Fatigue scale improvement (assessment of the level of discomfort caused by a state of fatigue)
Trail Making Test parts (A and B) | at weeks 12 and 52
  TMT test improvement
Improvement in Clinical Global Impression (CGI) | at weeks 12 and 52
  CGI improvement (patient progress and treatment response over time)
Aggregate Z-score of secondary endpoints. | at weeks 12 and 52
  Aggregate Z-score of secondary endpoints improvement

CONTACTS AND LOCATIONS:
Locations (6):
- Bulgaria (5):
  - Specialised Hospital for Active Treatment of pneumo-phthisiatric diseases - Burgas" EOOD, Pneumology ward, Burgas
  - Multiprofile Hospital for Active Treatment "Sv. Ivan Rilski" EOOD, Kozloduy
  - Multiprofile Hospital for Active Treatment "Sv. Paraskeva" OOD, Pleven
  - University Multiprofile Hospital for Active Treatment "Kaspela" EOOD Clinic of thoracic surgery, Plovdiv
  - University Multiprofile Hospital for Active Treatment "Aleksandrovska" EAD, Sofia
- Hospital of Skopje, Skopje, North Macedonia